CLINICAL TRIAL: NCT01260844
Title: An Open-Label Study to Evaluate the Effect of a Single Dose of Briakinumab on the Pharmacokinetics of Single Doses of Caffeine, Tolbutamide, Omeprazole, Metroprolol, and Midazolam in Subjects With Moderate to Severe Psoriasis
Brief Title: Open Label, Single Dose, Non-randomized Study to Assess the Drug to Drug Interaction of Briakinumab on CYP Substrates.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: M12-160
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-05

CONDITIONS: Moderate to Severe Plaque Psoriasis
MeSH Terms: interventions — briakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single dose of briakinumab (Experimental): single dose briakinumab cocktail of CYP substrates
  Interventions: Drug: briakinumab

INTERVENTIONS:
Drug: briakinumab — single dose briakinumab and 2 doses of CYP substrates
  Other Names: ABT-874 Briakinumab

SUMMARY:
Phase 1, drug-drug interaction study to evaluate the effects of Briakinumab on hte pharmacokinetics of single doses of CYP substrate in subjects with moderate to severe psoriasis.

DETAILED DESCRIPTION:
The study does involve 3 days confinement at the beginning of the trial and 4 days at the end of the trial. The trial duration is 17 days with 6 visits not including the confinement periods. The trial is being conducted in moderate to severe plaque psoriasis subjects. Serial blood samples will be taken after each doses of the CYP substrates are administered and blood samples will be collected for briakinumab PK and briakinumab ADA.

ELIGIBILITY:
Inclusion Criteria

1. Male or female and age is between 18 and 55 years, inclusive.
2. Clinical diagnosis of plaque psoriasis for at least 6 months as determined by subject's interview of his/her medical history and confirmation of diagnosis through physical examination by the investigator.
3. Moderate to severe plaque psoriasis defined by ≥ 10% Body Surface Area (BSA) involvement at the Screening visit and Day -2 visit.
4. PGA of at least moderate (defined as a PGA of ≥3) disease at the Screening visit and Day -2 visit.
5. Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, chest x-ray, and 12-lead electrocardiogram (ECG) performed at Screening.
6. Females must have negative results on all pregnancy tests during the study.
7. Body Mass Index (BMI) is between 18 to 29, inclusive.

Exclusion Criteria

1. History of either Type 1 or 2 diabetes
2. History of significant sensitivity to any drug
3. History of drug or alcohol abuse within 6 months prior to screening
4. Receipt of any investigational product within 1 month prior to day -2 , or current participation in any clinical study receiving any study drug or device
5. Use of known CYP inhibitors (e.g., ketoconazole, clotrimazole) or inducers (e.g., dexamethasone, phenytoin, rifampin, carbamazepine) within 1 month prior to Day -2
6. Use of known CYP substrates, (including hormonal contraception), within 1 month prior to Study Day-2. See Appendix E for List of Cytochrome P450 (CYP) Medications for the Treatment of Hypertension and Dyslipidemia
7. Receipt of any vaccine within 3 months prior to study drug administration
8. Subject has received vaccination with Bacille Calmette-Guérin (BCG)
9. Previous exposure to systemic anti-IL-12/23 therapy, including briakinumab (ABT-874) or ustekinumab.
10. Cannot discontinue systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis, during the study:

    * Non-biologic systemic (investigational or marketed) therapies must be discontinued at least 1 month prior to the Day-2
    * Biologic (investigational or marketed) therapies must be discontinued at least 12 weeks prior to Day-2
11. Subjects that must use topical therapies for the treatment of psoriasis such as corticosteroids, vitamin D analogs, or retinoids during the study. Subjects are allowed to use:

    * Shampoos that contain no corticosteroid;
    * Bland (without beta or alpha hydroxy acids) emollients;
    * Low potency (Class VI or Class VII) topical corticosteroids on the palms, soles, face, inframammary area, and groin only. See Appendix F for a Listing of Examples of Class VI and VII Topical Corticosteroids
12. Cannot avoid PUVA phototherapy during the study.
13. Subject is taking or requires oral, injectable or inhaled corticosteroids during the study.
14. Use of herbal or dietary supplements, such as St. John's Wort, within 1 month prior to Day -2 or 10 half lives whichever is longer.
15. Use of caffeine and/or theobromine (coffee, chocolate, tea, cola drinks, mountain dew etc.) within three days prior to Day-2 and Day 12.
16. Consumption of orange, grapefruit or orange or grapefruit products (juices), broccoli, brussels sprouts, or charcoal grilled meats within three days prior to Day-2 and Day 12
17. Consumption of alcohol within the 48 hours prior to Day-2 and Day 12.
18. Use of tobacco or nicotine-containing products within the 6-month period preceding Day-2.
19. Positive screen for drugs of abuse, alcohol or cotinine
20. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study or in the 60 days after receiving the single dose of study drug
21. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening, and the results will be maintained and communicated to the subjects confidentially by the study site.
22. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption
23. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks Day-2.
24. Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication exacerbated psoriasis, or new onset guttate psoriasis.
25. Poorly controlled medical condition, such as documented history of recurrent infections, unstable ischemic heart disease, congestive heart failure, recent cerebrovascular accidents and any other condition, or an unstable psychiatric condition which, in the opinion of the investigator and/or Abbott's Medical Monitor, would put the subject at risk by participation in the study
26. Subject has infection or risk factors for severe infections, for example:

    * Active tuberculous disease;
    * Evidence of latent tuberculosis (TB) infection demonstrated by a positive result of their Purified Protein Derivative (PPD) skin test
    * Subject is taking TB prophylaxis medication
    * Any other significant infection requiring hospitalization or intravenous (IV) antibiotics in the month prior to Day -2;
    * Infection requiring treatment with antibiotics in the month prior to Day -2
27. History of atherosclerotic cardiovascular disease as manifested by any of the following:
28. History of malignancies other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical carcinoma in situ
29. Exacerbation of asthma requiring hospitalization in the 10 years prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04

PRIMARY OUTCOMES:
Assessment of the drug-drug interaction potential of briakinumab (ABT-874) with cytochrome CYP 1A2. CYP2C9, CYP2C19, CYP2D6 and CYP3A4 in moderate to severe plaque psoriasis subjects | 17 days
  CYP Substrate cocktail administed at Day -1 and day 14 and Briakinumab at Day 1

SECONDARY OUTCOMES:
No secondary outcomes are reported for this study | No secondary outcomes are reported for this study
  No secondary outcomes are reported for this study

CONTACTS AND LOCATIONS:
Overall Officials: David A Williams, MD, Study Director — Abbott